CLINICAL TRIAL: NCT03037086
Title: A Retrospective Non-Interventional Study of PD-L1 Prevalence and Clinical Outcomes for Non-Small Cell Lung Cancer in Asia-Pacific
Brief Title: Asia PDL1 Study Among NSCLC Patients
Acronym: MEDI-APEX
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00002
Record Dates: First submitted 2016-10-05; First posted 2017-01-31 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Locally Advanced or Metastatic NSCLC
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumour tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One single cohort: One single cohort of NSCLC patients with disease diagnosis between January 2010 and December 2014. The locally advanced or metastatic NSCLC patients should have initiated 1st line palliative chemotherapy by end of 2014.

SUMMARY:
MEDI-APEX is a non-interventional, retrospective, cohort study to characterize PD-L1 expression and to assess the clinical characteristics and outcomes among NSCLC patients

DETAILED DESCRIPTION:
MEDI-APEX is a non-interventional, retrospective, cohort study to characterize PD-L1 expression among NSCLC patients and to assess the clinical characteristics and outcomes of these patients with specific attention to EGFR, ALK, and KRAS mutations. The study will determine whether PD-L1 is a prognostic factor in the Asia-Pacific patient population; The study will enrol NSCLC patients with disease diagnosis between January 2010 and December 2014; The patients will be recruited from Asia-Pacific, potentially China, Japan, and South Korea. A total of approximately 750 patients will be enrolled in the study; around 250 NSCLC patients will be enrolled per country.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female (according to age of majority as defined in local regulations).
2. NSCLC diagnosis between 01 January 2010 and 31 December 2014.
3. FFPET collected via core needle biopsy or resection and available in sufficient amount to complete PD-L1 testing.
4. FFPET tissue samples collected for NSCLC original diagnosis determination or for further analysis (e.g. research or treatment purposes) until the index date.
5. Patients with locally advanced or metastatic NSCLC who have initiated 1st line palliative chemotherapy by 31 December 2014.

Exclusion Criteria:

1. Patients with locally advanced NSCLC with resectable disease and treated with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with NSCLC, including SqCLC, diagnosed between 01 January 2010 and 31 December 2014
Sampling Method: Non-Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Characterization of PD-L1 expression among NSCLC patients | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
  Characterization of PD-L1 expression among locally advanced, unresectable NSCLC patients (Stage III) and newly diagnosed Stage IV or recurrent metastatic NSCLC patients.

SECONDARY OUTCOMES:
Examination of overall survival by PD-L1 status among NSCLC patients | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
Examination of disease-free survival (DFS) by PD-L1 status among NSCLC patients | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
Examination of relapse-free survival (RFS) by PD-L1 status among NSCLC patients | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
Examination of progression-free survival (PFS) by PD-L1 status among NSCLC patients | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
Description of patient characteristics by PD-L1 status among NSCLC patients. | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
Description of the overlap between PD-L1 expression and presence of EGFR, ALK or KRAS mutations among NSCLC patients | from NSCLC diagnosis date between January 2010 and December 2014 until index date, defined as the date of data abstraction
  And the prevalence of PD-L1 expression ≥25%, and ≥90%, will be calculated for each mutation status for the EGFR, ALK and KRAS biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-We Kim, Prof., Principal Investigator — Asan Medical Center; Hiroyuki Suzuki, Dr., Principal Investigator — Fukushima Medical University Hospital; Noriyuki Ebi, Dr., Principal Investigator — Aso Co.,Ltd Iizuka Hospital; Li Zhang, Prof., Principal Investigator — Sun Yat-sen University; Ping Yu, Prof., Principal Investigator — Sichuan Province Cancer Hospital
Locations (4):
- Research Site, Guangzhou, Guangdong, China
- Japan (2):
  - Research Site, Iizuka-shi, Fukuoka
  - Research Site, Fukushima, Fukushima
- Research Site, Seoul, South Korea

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3870&filename=D4191R00002_Synopsis_Redacted.pdf